CLINICAL TRIAL: NCT04863820
Title: Small Peripheral Fibers Assessment Using Cutaneous Silent Period In Normal Individuals In Egypt
Brief Title: Small Fiber Assessment by Cutaneous Silent Period
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sarah Mostafa Kaddah, Clinical Neurophysiology resident, Cairo University
Other Study IDs: Clinical Neurophysiology
Record Dates: First submitted 2021-04-14; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Small Fiber Neuropathy
MeSH Terms: conditions — Small Fiber Neuropathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: cutaneous silent period — form of Nerve conduction studies

SUMMARY:
Our primary objective in this study is to investigate the cutaneous silent period (CSP) in normal subjects in the Egyptian population, as it was not carried out before in Egypt. The aim was to carry out the test in our unit to study the appropriate method, technique, and parameters of this new test so that we can apply it in future research. In addition, to obtain preliminary normative data of the test; onset latency, end latency, duration, and latency difference (LD) of CSP, as well as assess the effect of age, height, upper limb length, and gender on CSP values.

DETAILED DESCRIPTION:
Nerve conduction studies performed routinely in electromyoneurography laboratories deal mainly with large myelinated fast conducting nerve fibers. A reliable method allowing the study of small peripheral nerve fibers (Aδ & C) would be of interest (Jovita et al., 2006). As they are initially affected and maybe the earliest exhibited sign of neuropathy.

In recent years, the cutaneous silent period (CSP) has received increased attention in health and disease. The CSP is an inhibitory spinal reflex that appears following strong electrical stimulation of the cutaneous nerve and causes suppression of voluntary muscular contraction for a certain period of time (Kofler et al., 2019). This action presents a reciprocal action to the nociceptive flexor withdrawal response (FWR) which serves as an 'excitatory reflex' increasing activity in primary flexor muscles. When taken into context, the interplay between the CSP and FWR can clearly be seen.

The evaluation of the CSP represents a useful electrophysiological method for investigating the function of small fibers by using standard electromyography equipment (Eckert et al., 2018).

ELIGIBILITY:
Inclusion criteria:

* Healthy participants able to cooperate and to follow instructions.
* Participants having a normal value for electrophysiological parameters (Nerve conduction studies)
* Participants must be free from any musculoskeletal impairment of the limbs

Exclusion criteria:

* Participants with neurological disorders
* Participants with cognitive impairment
* Participants receiving medications that may affect the NCS
* Participants with small fiber neuropathy (burning sensation, pricking sensation, allodynia, and hyperalgesia)
* Participants with an abnormal value for Nerve conduction studies
* Participants with musculoskeletal impairment of the limbs

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Gender: males and females, age group: 20-60, healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2021-04-27 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Normative parameters of cutaneous silent period of the median, ulnar , and sural nerves (measured in milli second) | 1 year
  establishing Normative of CSP enables the diagnosis of small fiber neuriopathy in the future The CSP parameters include: CSP onset latency,CSP end latency, and CSP duration (measured in ms; milli second)

CONTACTS AND LOCATIONS:
Overall Officials: Hebatallah R Rashad, Professor, Study Director — Cairo University; Lamia M Afifi, Professor, Study Director — Cairo University; AlShaimaa S Khalil, MD, Study Director — Cairo University
Locations (1):
- Medicine, Cairo, Egypt

REFERENCES:
- [Background] Svilpauskaite J, Truffert A, Vaiciene N, Magistris MR. Electrophysiology of small peripheral nerve fibers in man. A study using the cutaneous silent period. Medicina (Kaunas). 2006;42(4):300-13. PMID 16687902
- [Background] Onal MR, Ulas UH, Oz O, Bek VS, Yucel M, Taslipinar A, Odabasi Z. Cutaneous silent period changes in Type 2 diabetes mellitus patients with small fiber neuropathy. Clin Neurophysiol. 2010 May;121(5):714-8. doi: 10.1016/j.clinph.2009.12.024. Epub 2010 Feb 6. PMID 20138004
- [Background] Lopergolo D, Isak B, Gabriele M, Onesti E, Ceccanti M, Capua G, Fionda L, Biasiotta A, Di Stefano G, La Cesa S, Frasca V, Inghilleri M. Cutaneous silent period recordings in demyelinating and axonal polyneuropathies. Clin Neurophysiol. 2015 Sep;126(9):1780-9. doi: 10.1016/j.clinph.2014.11.013. Epub 2014 Nov 25. PMID 25497713
- [Background] Eckert NR, Poston B, Riley ZA. Differential processing of nociceptive input within upper limb muscles. PLoS One. 2018 Apr 25;13(4):e0196129. doi: 10.1371/journal.pone.0196129. eCollection 2018. PMID 29694394